CLINICAL TRIAL: NCT04417374
Title: Caracteristics of the Patients Hospitalized With Unvonluntary Commitment Procedure, in Pandemic and Confinement Context
Brief Title: Caracteristics of the Patients Hospitalized With Unvonluntary Commitment Procedure, in the Context COVID-19
Acronym: HoCoPsy
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0320
Record Dates: First submitted 2020-06-03; First posted 2020-06-04 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: COVID 19; Disease Outbreak; Mental Disorders
Keywords: Confinement; Disease outbreak; Unvonluntary commitment
MeSH Terms: conditions — COVID-19; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unvonluntary commitment from March 12th to April 09th 2019: Patients hospitalized with unvonluntary commitment procedure from March 12th to April 09th 2019
  Interventions: Other: Description of groups caracteristics
- Unvonluntary commitment from March 12th to April 09th 2020: Patients hospitalized with unvonluntary commitment procedure from March 12th to April 09th 2020
  Interventions: Other: Description of groups caracteristics

INTERVENTIONS:
Other: Description of groups caracteristics — Comparison of the two groups on all the following criterias : age, sex, if the patient lives alone, the matter of hospitalization, its lengh, their primary psychiatric diagnostic, the use of toxics at the moment of the hospitalization and if this psychiatric decompensation happens in a context of treatment interruption.

SUMMARY:
The actual worldwide context (disease outbreak, confinements instaured in many countries) is a stressful factor for many people. It can have consequences on mental health : separation from loved ones, loss of freedom, uncertainty about infection status, boredom. Patients with mental disorders are especially vulnerable.

On march 17th, the french government ordonned a national confinement to slow the progression of the COVID-19 outbreak, for 15 days at first then renewed several times. This situation has led to a reorganization of care as requested on March 22nd, 2020 in the recommendations applicable to the organization of care in psychiatric services : priority to telephone contacts and teleconsultation by multiplying contacts and assessments.

By the time the reorganization of care became operational, the most vulnerable patients may have experienced a decompensation of their disease.

It is important to know if the COVID-19 outbreak combined with the confinement increased the number of unvoluntary commitment the month after the announce of the confinement.

This could help us understand which patients are more vulnerable is this context, and improve our organization (ambulatory and hospitalization care) if this situation occurs again.

DETAILED DESCRIPTION:
The main objective is to notice if we can observe a increase in the number of unvonluntary commitment the month after the announce of the confinement in the psychiatric hospital La Colombière, CHU Montpellier, France.

Secondary objectives :

* Describe the causes of unvonluntary commitment, and the principal psychiatric diagnostic of the patients
* Assess the lengh of the hospitalization
* Assess the number of patients hospitalized without psychiatric antecedent
* Assess the number of treatment interruptions in the recent history before hospitalization
* Asses the number of patients living alone
* Asses the number of patients using drugs

It is expected to highlight :

* An increase of the number of unvontuntary commitment
* If one or several mental disorders were more at risk of requiring an unvonluntary commitment
* An increased lengh of hospitalization
* An increased number of unvonluntary commitment of patients without psychiatric antecedent
* An increased number of treatment interruptions
* A link between hospitalization and living alone
* A link between hospitalization and using drugs

The medical file of all the patients unvonlutary commited from march 12th to April 09th 2020 are screened, and compared to the patients unvonlutary commited during the same period in 2019.

The caracteristics of interest are their age and sex, if the patient lives alone, the matter of hospitalization, its lengh, their primary psychiatric diagnostic, the use of toxics at the moment of the hospitalization and if this psychiatric decompensation happens in a context of treatment interruption.

ELIGIBILITY:
Inclusion criteria:

- Unvonluntary commitment in psychiatric hospital La Colombière, CHU Montpellier, from march 12th to april 19th (2019 and 2020).

Exclusion criteria:

- refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults having been aditted to the psychiatric hospital La Colombière, CHU Montpellier, France, with unvonluntary commitment procedure from march 12th to April 09th (2019 and 2020)
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number of hospitalized patients | 1 months
  Number of hospitalized patients From March 12th to April 09th

SECONDARY OUTCOMES:
Cause of hospitalization | 1 months
  Primary psychiatric diagnostic From March 12th to April 09th

OTHER OUTCOMES:
Lengh of hospitalization | 1 months
  Patients without psychiatric antecedent (number) From March 12th to April 09th
Treatment interruption | 1 months
  Presence of absence of history of treatment interruption leading to the hospitalization From March 12th to April 09th
Number of hospitalized patients living alone | 1 months
  Number of hospitalized patients living alone (opposed to those living with family) From March 12th to April 09th
Use of drugs | 1 months
  Number of patients using drugs From March 12th to April 09th

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Olie, MD PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC